CLINICAL TRIAL: NCT04485455
Title: Open Label Study of the Efficacy, Durability, Safety and Feasibility of Intermittent Theta Burst Stimulation (iTBS) in Adolescents With Major Depressive Disorder: Effect Duration, Suicidality, and Non-Suicidal Self Injurious Behavior
Brief Title: iTBS for Adolescent Depression: An Open Label Study Evaluating Safety and Efficacy of Treatment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 19-1100
Record Dates: First submitted 2020-07-21; First posted 2020-07-24 (Actual); Results first posted 2021-11-30 (Actual); Last update posted 2021-11-30 (Actual); Status verified 2021-11

CONDITIONS: Depression
Keywords: Adolescent Depression; Teen Depression
MeSH Terms: conditions — Depression

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- iTBS Therapy (Experimental): Teenage participants with depression will receive iTBS therapy using a Transcranial Magnetic Stimulation (TMS) protocol delivering electro-magnetic stimulation
  Interventions: Device: iTBS Device/Motor Threshold Coil; Device: iTBS Device/Treatment Coil

INTERVENTIONS:
Device: iTBS Device/Motor Threshold Coil — Motor Threshold determination, done prior to starting treatments, determines the location and the intensity for the iTBS treatments. A magnetic field is applied with increasing intensity stimulating the motor region of the brain until there is thumb movement; this indicates the intensity of the treatments; the location for treatment is in the sensory area parallel to this location.
  Other Names: MagProX100 with MagOption Stimulator and Magpro Coil C-B60 or C-B70
Device: iTBS Device/Treatment Coil — iTBS is a particular TMS protocol which delivers the magnetic field in triplet bursts (three stimulations very close together at a frequency of 50 Hz very quickly). The triplet bursts are repeated at a rate of 5 Hz for 2 seconds (30 pulses), followed by 8 seconds rest, repeated 20 times for a total of 600 pulses. Each treatments lasts approximately 3 minutes, and sessions are provided 20 times (Monday-Friday for 4 consecutive weeks).
  Other Names: MagPro, Models R30 with MagOption, X100 WITH MagOption, Coil Cool-B65

SUMMARY:
This is an open label, pilot, feasibility study evaluating effects of Intermittent Theta Burst Transcranial Magnetic Stimulation (iTBS) on 5 eligible adolescents for the treatment of depression. Safety and tolerability will be evaluated with changes in depression scores, and suicidality and non-suicidal self injurious behavior will also be monitored for exploratory and safety measures.

DETAILED DESCRIPTION:
This study will investigate the efficacy and durability of the effects of Intermittent Theta Burst Stimulation (iTBS) in adolescent depression by measuring changes in clinical ratings before, during, and after 4 weeks of treatment, up to 12 weeks following treatment. The investigators expect that subjects will show: improvement in symptoms over 20 iTBS sessions as measured by the Children's Depression Rating Scale Revised (CDRS-R), Hamilton Depression Rating Scale (HAM-D) and Non-suicidal Self Injurious Behavior (NSSIB) measures, and persistence of this reduction of depressive symptoms through the 12 weeks follow up period of the study. In this study, the investigators will investigate the safety of the effects of iTBS in adolescent depression. The investigators will investigate safety of the treatment regimen by assessing suicidality. The investigators expect suicidal thoughts and behavior will reduce with iTBS treatment as measured by the Columbia Suicide Severity Rating Scale (C-SSRS) and a psychiatrist's clinical assessment. The investigators also expect that those with NSSIB at the start of the trial will have less after iTBS treatments. The investigators do not expect any change in cognition measured with the Mini Mental Status Exam (MMSE), Trails B, and List Generation. The investigators will investigate treatment feasibility by assessing treatment completion and withdrawal. The investigators define the feasibility of iTBS will be defined as feasible by as completion of 15/20 (75%) iTBS treatment sessions by all subjects and withdrawal from treatment of no more than one of five subjects (20%) due to intolerable side effects or persistent symptoms of MDD. Investigation of efficacy, durability, safety as well as feasibility simultaneously is essential in this preliminary study of the use of iTBS in adolescents in order to justify a larger future study. This study will include a screening visit, 20 iTBS treatments, and 3 planned follow up visits.

ELIGIBILITY:
Inclusion Criteria:

* A score of greater than 40 on the CDRS-R and 17 on HAM-D.
* Documentation of DSM-V criteria for current MDD or TRD will be required for study entry.
* Patients may be on antidepressant medication at a stable dose or receiving psychotherapy with a licensed provider during the active phase of TMS treatment for 4 weeks.
* Ability to provide consent and take part in questionnaires and scales (i.e.: not currently intellectually disabled).
* The presence of suicidality or NSSIB are not required to enter this study. Although our secondary end-points include suicidality, and the investigators are also exploring NSSIB, and thus this may not lead to many data, the investigators' plan is to use data from this study to justify a larger study where this can be more robustly investigated.

Exclusion Criteria:

* Past or current diagnosis of bipolar disorder, psychosis, seizures or traumatic brain injury.
* Presence of intracranial metallic implants or fragments, which is a contraindication for TMS.
* Lifetime history of (or currently present) epilepsy.
* Current diagnosis of substance abuse, eating disorder, PTSD (Post Traumatic Stress Disorder), or intellectual disability.* Nicotine use disorder will not directly preclude a potential subject from this study. Although chronic nicotine use does effect central nervous system excitability, what would be more confounding to our study would be if there is a sudden change in nicotine use during the treatment phase, as this may affect the motor threshold. Inclusion will however be at the PI's discretion.
* Current imminent suicide ideation or other clinical reasons for inpatient psychiatric hospitalization.
* Currently pregnant. There is currently not adequate data from this population to ensure safety with the scope of this protocol.
* Any reason the investigator determines may cause noncompliance with study rules or is unfit for receiving treatment.
* Currently taking certain medications including antidepressants, stimulants, benzodiazepines, and antipsychotics, antiepileptic (per investigator discretion).
* Any positive drug testing from a urine drug test unless medically indicated with a valid prescription.

  * Those with marijuana/cannabis positive results may retest later if at that time they do not meet criteria for substance abuse at screening and agree to refrain from use for the duration of study participation. Decision to be made by Investigator discretion.

Ages: 13 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 5 (Actual)
Dates: Start 2020-09-21 (Actual); Primary Completion 2021-04-30 (Actual); Study Completion 2021-07-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Shahzad Ali, MD, Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- University of North Carolina at Chapel Hill-Psychiatry Outpatient Clinic, Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Yes
Deidentified individual data that supports the results will be shared beginning 9 to 36 months following publication provided the investigator who proposes to use the data has approval from an Institutional Review Board (IRB), Independent Ethics Committee (IEC), or Research Ethics Board (REB), as applicable, and executes a data use/sharing agreement with UNC.
Supporting Information: Study Protocol, ICF
Time Frame: 9 to 36 months following publication
Access Criteria: Approval from an IRB, IEC, or REB and an executed data use/sharing agreement with UNC.

RESULTS

PARTICIPANT FLOW:
Groups:
- iTBS Open Label: All subjects enrolled into this study were in the same group, with all receiving active Intermittent Theta Burst Stimulation (iTBS) treatment.
Period: Overall Study
Arm/Group | iTBS Open Label
Started | 5
Completed | 5
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- iTBS Open Label: All subjects enrolled into this study were in the same group, with all receiving active iTBS treatment.
Arm/Group | iTBS Open Label
Number analyzed (Participants) | 5
Age, Continuous [Mean (Full Range); unit: years]
  13 to 17 year old | 16.2 [13 to 17]
Age, Customized [Count of Participants; unit: Participants]
  Age 17 | 4
  Age 13 | 1
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Female | 2
  Male | 2
  Non-Binary | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 1
  Unknown or Not Reported | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 4
  More than one race | 1
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 5
Mean Depression HAM-D Rating Score [Mean (Full Range); unit: Score on scale] — Depression rating is determined by (Hamilton Depression Rating Scale) HAM-D assessments. A higher score indicates more severe depression rating. Scores can range from 0-52.
  Score on scale | 16.8 [8 to 29]
Mean Depression CDRS-R Rating Score [Mean (Full Range); unit: Score on an assessment] — Depression rating is determined by Children's Depression Rating Score Revised (CDRS-R) assessments. A higher score indicates more severe depression rating. Scores for this assessment range from 17-113.
  Score on an assessment | 65.2 [50 to 75]

OUTCOME MEASURES:

1. Primary Outcome: Change in HAM-D Score From Baseline to Week 1
Description: The Hamilton Rating Scale for Depression (HAM-D) total score comprises a sum of the 17 individual item scores which ranges from 0 to 52. Higher scores indicate a greater degree of depression.
Time Frame: Baseline, Week 1
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | iTBS Open Label
Number analyzed (Participants) | 5
score on a scale | -7.6 [-15 to -0.42]

2. Primary Outcome: Change in CDRS-R Score From Baseline to Week 1
Description: The Children's Depression Rating Scale-Revised (CDRS-R) total score ranges from 17 (minimal or no symptoms of depression) to 113 (indicative of depression) is a semi-structured, clinician-rated instrument designed for use with children and adolescents between the ages of 6 to 17 years of age and their caregivers. The CDRS-R evaluates the presence and severity of symptoms commonly associated with depression in childhood.
Time Frame: Baseline, Week 1
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | iTBS Open Label
Number analyzed (Participants) | 5
score on a scale | -9.0 [-15 to -3.5]

3. Primary Outcome: Change in HAM-D Score From Baseline to Week 2
Description: as for outcome 1
Time Frame: Baseline, Week 2
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | iTBS Open Label
Number analyzed (Participants) | 5
score on a scale | -6.2 [-13 to 0.44]

4. Primary Outcome: Change in CDRS-R Score From Baseline to Week 2
Description: as for outcome 2
Time Frame: Baseline, Week 2
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | iTBS Open Label
Number analyzed (Participants) | 5
score on a scale | -16 [-24 to -7.5]

5. Primary Outcome: Change in HAM-D Score From Baseline to Week 3
Description: as for outcome 1
Time Frame: Baseline, Week 3
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | iTBS Open Label
Number analyzed (Participants) | 5
score on a scale | -9.2 [-15 to -3.5]

6. Primary Outcome: Change in CDRS-R Score From Baseline to Week 3
Description: as for outcome 2
Time Frame: Baseline, Week 3
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | iTBS Open Label
Number analyzed (Participants) | 5
score on a scale | -11 [-22 to -0.07]

7. Primary Outcome: Change in HAM-D Score From Baseline to Week 4
Description: as for outcome 1
Time Frame: Baseline, Week 4
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | iTBS Open Label
Number analyzed (Participants) | 5
score on a scale | -7.8 [-14 to -1.6]

8. Primary Outcome: Change in CDRS-R Score From Baseline to Week 4
Description: as for outcome 2
Time Frame: Baseline, Week 4
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | iTBS Open Label
Number analyzed (Participants) | 5
score on a scale | -14 [-23 to -4.3]

9. Secondary Outcome: Number of Occurrences of Passive Suicidal Ideation
Description: Columbia Suicide Severity Rating Scale (C-SSRS) is a semi-structured interview that has "yes or no" answers to assess the likelihood of a subject harming themselves, including "yes/no" to passive suicidal ideation. Participants indicating a "yes" response to any of these questions were reported as having passive suicidal ideation. Each participant was assessed at 8 timepoints during the study.
Time Frame: Up to 12 Weeks Post-Treatment Completion, a total of up to 16 weeks
Measure: Number; unit: Occurrences passive suicidal ideation
Arm/Group | iTBS Open Label
Number analyzed (Participants) | 5
Occurrences passive suicidal ideation
  Baseline | 2
  Treatment Week 1 | 2
  Treatment Week 2 | 1
  Treatment Week 3 | 0
  Treatment Week 4 | 2
  Follow Up Week 1 | 2
  Follow Up Week 4 | 0
  Follow Up Week 12 | 1

10. Secondary Outcome: Number of Participants Who Completed the Study
Description: Feasibility for this protocol is partially determined by completion rate. Treatment completion is defined in this protocol by 75% of treatments completed (15/20) per subject. This will be measured through completion of Week 4 of treatment (Week 5 of protocol when including screening phase).
Time Frame: Up to Week 5
Measure: Count of Participants; unit: Participants
Arm/Group | iTBS Open Label
Number analyzed (Participants) | 5
Participants | 5

11. Secondary Outcome: Number of Participants Who Withdrew From the Study
Description: Feasibility for this protocol is partially determined by withdrawal rate. Withdrawal is defined as no more than 1 out of 5 subjects (20% of participants) withdrawing due to intolerable side effects caused by treatment or persistent depressive symptoms. This will be measured through completion of Week 4 of treatment (Week 5 of protocol when including screening phase).
Time Frame: Up to Week 5
Measure: Count of Participants; unit: Participants
Arm/Group | iTBS Open Label
Number analyzed (Participants) | 5
Participants | 0

12. Secondary Outcome: Durability of Treatment Effect With HAM-D Scores
Description: Change in scores of Hamilton Depression Rating Scale (HAM-D) will be evaluated comparing Baseline to each follow-up phase at 1 week, 4 weeks, and 12 weeks post-treatment. The (HAM-D) total score comprises a sum of the 17 individual item scores which ranges from 0 to 52. Higher scores indicate a greater degree of depression.
Time Frame: From Baseline up to 12 Weeks Post-Treatment Completion, a total of up to 16 weeks
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | iTBS Open Label
Number analyzed (Participants) | 5
score on a scale
  Follow Up Week 1 | -8.8 [-14 to -3.2]
  Follow Up Week 4 | -11 [-17 to -3.8]
  Follow Up Week 12 | -9.4 [-15 to -4.2]

13. Secondary Outcome: Durability of Treatment Effect With CDRS-R Scores
Description: Change in scores of Children Depression Rating Scale Revised (CDRS-R) during follow-up phase at 1 week, 4 weeks, and 12 weeks post-treatment. The Children's Depression Rating Scale-Revised (CDRS-R) total score ranges from 17 (minimal or no symptoms of depression) to 113 (indicative of depression) is a semi-structured, clinician-rated instrument designed for use with children and adolescents between the ages of 6 to 17 years of age and their caregivers. The CDRS-R evaluates the presence and severity of symptoms commonly associated with depression in childhood.
Time Frame: Up to 12 Weeks Post-Treatment Completion, a total of up to 16 weeks
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | iTBS Open Label
Number analyzed (Participants) | 5
score on a scale
  Follow Up Week 1 | -21 [-33 to -7.9]
  Follow Up Week 4 | -19 [-32 to -6.2]
  Follow Up Week 12 | -23 [-34 to -12]

14. Secondary Outcome: Number of Occurrences of Non-Suicidal Self Injurious Behavior Through SITBI
Description: Self Injurious Thoughts and Behavior Interview (SITBI) is a semi-structured interview commonly used and administered by a clinician to determine if self-harm behavior has been present since the last visit. This will be evaluated at baseline (screening), once per week during the treatment phase, and at each follow up visit.
Time Frame: Up to 12 Weeks Post-Treatment Completion, a total of up to 16 weeks
Measure: Number; unit: Occurrences self-harm behavior
Arm/Group | iTBS Open Label
Number analyzed (Participants) | 5
Occurrences self-harm behavior
  Baseline | 0
  Treatment Week 1 | 0
  Treatment Week 2 | 0
  Treatment Week 3 | 0
  Treatment Week 4 | 0
  Follow Up Week 1 | 0
  Follow Up Week 4 | 0
  Follow Up Week 12 | 0

ADVERSE EVENTS:
Time Frame: From date of informed consent to completion of study, which is the last follow-up visit, an approximate total of 16 weeks.
Arm/Group | iTBS Open Label
All-Cause Mortality (participants affected / at risk) | 0/5
Serious Adverse Events (participants affected / at risk) | 0/5
Other Adverse Events (participants affected / at risk) | 5/5
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | iTBS Open Label (N=5)
Scalp Pain - mild (Musculoskeletal and connective tissue disorders) | 3 (8)
Scalp Pain - moderate (Musculoskeletal and connective tissue disorders) | 3 (3)
Ear Pain - mild (Musculoskeletal and connective tissue disorders) | 1 (1)
Jaw Twitching - mild (Musculoskeletal and connective tissue disorders) | 5 (12)
Jaw Twitching - moderate (Musculoskeletal and connective tissue disorders) | 2 (2)
Tingling (Musculoskeletal and connective tissue disorders) | 1 (1)
Right arm twitch - moderate (Musculoskeletal and connective tissue disorders) | 1 (1)
Right arm twitch - mild (Musculoskeletal and connective tissue disorders) | 2 (3)
Burn on shoulder - moderate (Skin and subcutaneous tissue disorders) | 1 (1)
Fever - mild (Immune system disorders) | 1 (1)
Anxiety in social setting - mild (Psychiatric disorders) | 1 (1)
Eyebrow twitching - mild (Musculoskeletal and connective tissue disorders) | 3 (9)
Eye twitching - moderate (Musculoskeletal and connective tissue disorders) | 1 (3)
Migraine - severe (Nervous system disorders) | 1 (1)
Headache - mild (Nervous system disorders) | 1 (2)
Headache- moderate (Nervous system disorders) | 1 (2)
Arm soreness - moderate (Musculoskeletal and connective tissue disorders) | 1 (2)
Arm soreness - mild (Musculoskeletal and connective tissue disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-12-03): https://cdn.clinicaltrials.gov/large-docs/55/NCT04485455/Prot_SAP_000.pdf
  • Informed Consent Form (2020-09-29): https://cdn.clinicaltrials.gov/large-docs/55/NCT04485455/ICF_001.pdf